CLINICAL TRIAL: NCT02330484
Title: Affect of Incentive Strategy on the Adherence to Medication Among Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCEMD-026
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: Community management， incentives, Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- incentives to physicians (Experimental): Give incentives to physicians according to patients' HbA1c improvement
  Interventions: Behavioral: Give incentives to physician based on their patient's HbA1c improvement
- incentives to patients (Experimental): Give incentives to patients according to their HbA1c improvement
  Interventions: Behavioral: Give incentives to patients based on their own HbA1c improvement
- incentives to both physicians and patients (Experimental): intervention mode: Give incentives to physicians and patients according to patients' HbA1c improvement
  Interventions: Behavioral: Give incentives to patients based on their own HbA1c improvement; Behavioral: Give incentives to physician based on their patient's HbA1c improvement
- Group with no incentives (No Intervention)

INTERVENTIONS:
Behavioral: Give incentives to patients based on their own HbA1c improvement — Give incentives to patients based on their own HbA1c improvement
  Arms: incentives to both physicians and patients; incentives to patients
Behavioral: Give incentives to physician based on their patient's HbA1c improvement — Give incentives to physician based on their patient's HbA1c improvement
  Arms: incentives to both physicians and patients; incentives to physicians

SUMMARY:
Based on patients' HbA1c improvement, this study aims to establish an incentive strategy to family physicians and patients respectively to evaluate the affect on the adherence to medication among patients with type2 diabetes.

DETAILED DESCRIPTION:
First step: In this study, the investigators will conduct an open-label controlled randomized cluster trial to enroll 400 eligible and voluntary patients with type 2 diabetes from the community. 16 physicians will be involved in this study for patient management. Each physician will care at least 20 patients as a random unit which will be divided into 4 groups for baseline assessment including demographic characteristics, diabetes diagnosis and treatment, complication, biochemical indexes and self-management. The involved patients and physicians will receive related training. The patients will sign the informed consent form.

Second step: This study aims to give incentives to physicians or patients or both the physicians and patients based on HbA1c improvement. All the patients will sign the informed consent form. Regarding to the control group, health courses and community management will be given as usual. the investigators will evaluate the condition of patients' medication adherence after giving the incentives.

Third step: MEMS will be used in the intervention to monitoring patients' medication adherence. As a monitoring instrument, MEMS (Aardex, Zurich, Switzerland) is a plastic container with a spring-loaded device in the cap. Each time the bottles is opened for at least 3 seconds, the time and date of opening are recorded and saved. Based on the research data and the HbA1c improvement, this study will analyze the other factors which affect the patients' adherence to medication. Meanwhile, the investigators will collect patients' information such as blood pressure, biochemical index, complications related to diabetes, life quality, self-management, life style, health behavior, medications, health expenditure so as to evaluate the affect of incentive strategy on the adherence to medication among patients with type 2 diabetes.

Endpoint of the study:

The study will be ended in 12 months, endpoint measurement indicators are listed below:

1. The study will be ended in 12 months
2. Patient's drop out of the study
3. Stopping taking oral hypoglycemic drugs
4. The diabetic condition worsen, needs surgery or hospitalization treatment
5. Frequency of severe hypoglycemia or other complications that can not continue the study
6. Death of the patient

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed type 2 diabetes patients (ICD9) according to the medical record and patient's disease history
2. 40 to 74 years old
3. Diagnosis type 2 diabetes more than 6 months
4. Take at least one kind of oral hypoglycemic medication(including insulin injection)
5. Got treatment in community hospitals or follow up for more than 12 months
6. Have medical insurance
7. Stable condition with no adverse indication
8. Participate in this study voluntarily and sign the inform consent from

Exclusion Criteria:

1. Terminal illness
2. Serious hearing and visual disorder
3. Intend to receive selective surgery, to get pregnancy and breast feeding in three months
4. Demnentia or communication disorders
5. Mental disorders
6. The paralyzed or the handicapped
7. Expected survival time less than one-year

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemic Medication adherence rates using electronically monitored adherence (MEMS cap) data | 12 months
  MEMS will be used in the intervention to monitoring patients' medication adherence. As a monitoring instrument, MEMS (Aardex, Zurich, Switzerland) is a plastic container with a spring-loaded device in the cap. Each time the bottles is opened for at least 3 seconds, the time and date of opening are recorded and saved.

SECONDARY OUTCOMES:
Self-report medication adherence | 12 months
  The investigators assess adherence with MMAS 8-item version and BMQ-specific.
Improvement of HbA1c | 12 months
Score on the Diabetes Quality Of Life | 12 months
MEMS cap data compared to PHQ-9 and AIS assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liebin Zhao, MSM, Study Chair — Shanghai Clinical Centre for Endocrinology and Metabolism
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China